CLINICAL TRIAL: NCT02519816
Title: Continuous Alloreactive T Cell Depletion and Regulatory T Cell Expansion for the Treatment of Steroid-refractory or Dependent Chronic GVHD
Acronym: CARE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: daphne brockington (Other)
Responsible Party: Sponsor-Investigator, daphne brockington, Dr. Imran Ahmad, Maisonneuve-Rosemont Hospital
Organization: Maisonneuve-Rosemont Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CNTRP 1401
Record Dates: First submitted 2015-07-16; First posted 2015-08-11 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic GVHD After HCT for Cancer or Immune Disease
Keywords: post stem cell transplantation; Steroid refractory; dependent chronic
MeSH Terms: conditions — Immune System Diseases | interventions — Dimethyl Sulfoxide; Plasmalyte A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Open-label phase II study. After signing informed consent, patients will undergo 6 times an apheresis during the 6-month treatment period. These cells will be manufactured into the Rhitol and frozen in aliquots. Then re-infused.
  Interventions: Other: Autologous peripheral blood mononuclear cells ex vivo depleted for reactive T cells, using TH9402 based photodynamic therapy, in a final formulation of 10% DMSO, 30% autologous plasma in PlasmaLyte.

INTERVENTIONS:
Other: Autologous peripheral blood mononuclear cells ex vivo depleted for reactive T cells, using TH9402 based photodynamic therapy, in a final formulation of 10% DMSO, 30% autologous plasma in PlasmaLyte.

SUMMARY:
Phase II multicenter, Canadian only study - open to 25 subjects. Study open to subjects with steroid-refractory or dependent chronic graft vs host disease.

Series of 6 aphereses and 28 re-infusions over 24 weeks. Primary endpoint is FFS at 24 weeks. Primary objective is to measure the efficacy of CARE (Continuous Alloreactive T-Cell depletion and Regulatory T-cell Expansion)

ELIGIBILITY:
Inclusion Criteria: (Main)

* 1. Newly diagnosed chronic GVHD as defined by the National Institutes of Health (NIH) Consensus with no more than 24 weeks of treatment with systemic steroids.

AND 2. Chronic GVHD must be refractory or dependent to standard therapy, defined as (one of the following):

* Progression on prednisone 7 mg/kg/week for 2 weeks, or
* Stable disease on ≥ 3.5 mg/kg/week of prednisone for 4-8 weeks, or
* Inability to taper prednisone below 3.5 mg/kg/week.

Exclusion Criteria: (Main)

* 1. Persistent, recurrent or late-onset acute GVHD, without signs of chronic GVHD.

OR 2. Overlap GVHD syndrome with uncontrolled features of previously diagnosed acute GVHD.

OR 3. Treatment with more than two systemic non-steroidal immunosuppressants within 4 weeks prior to enrollment.

OR 4. Time from allogeneic transplantation > 2 years. OR 5. Lymphocyte count < 0.2 x 109/L on two last consecutive CBCs before inclusion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03; Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is failure-free survival (FFS) at 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Maissoneuve, Montreal, Quebec, Canada